CLINICAL TRIAL: NCT02515123
Title: Promotion of Regular Oesophageal Motility to Prevent Regurgitation and Enhance Nutrition Intake in Long-stay ICU Patients. A Multicenter, Phase II, Sham-controlled, Randomized Trial. The PROPEL Study
Brief Title: Promotion of Oesophageal Motility to Prevent Regurgitation and Enhance Nutrition Intake in ICU Patients.
Acronym: PROPEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: E-Motion Medical Ltd. (Industry)
Collaborators: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROPEL (ICU-02)
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Critically Ill; Malnutrition
Keywords: intensive care unit; malnutrition; GI motility; nutritional intake
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E-Motion System (Experimental): E-motion tube + E-motion EPG 1000
  Interventions: Device: E-Motion System
- E-Motion Sham Decive (Sham Comparator): E-motion tube + SHAM E-motion EPG 1000
  Interventions: Device: Sham E-Motion System

INTERVENTIONS:
Device: E-Motion System — E-Motion Tube: A disposable oro/nasogastric feeding tube fitted with stainless steel electrodes along its length that delivers the stimulation to the esophageal mucosa.
  E-motion EPG 1000: a durable, touchscreen operated, bedside control unit that generates the electric stimulation pattern and sends it via the feeding tube to the esophagus.
  By applying predetermined sequences of electrical stimulation to various locations along the esophagus asynchronous esophageal motion is induced, resulting is reduction of reflux and increased GI motility, enabling safer and better feeding.
  Arms: E-Motion System
Device: Sham E-Motion System — The sham EPG will resemble the investigational EPG. The external shape, interface, lights, and switches will be exactly the same. The Sham device will emit a low intensity pulsation so that, it will not unblind the patient nor health care professional. In the event that unblinding does occur, we will take steps to mask the identity of the EPG by covering the number of the device with tape to prevent members of the clinical team becoming aware of which device is active or sham.
  Arms: E-Motion Sham Decive

SUMMARY:
Early enteral feeding is a key component of the management of critically ill patients receiving mechanical ventilation. However, enteral feeding has been associated with serious complications such as gastro-esophageal reflux, with both overt and micro pulmonary aspiration, which potentially increases the risk to nosocomial pneumonia. Many critically ill patients experience poor tolerance of early enteral nutrition because of impaired gastric motility, which leads to a sequence of delayed gastric emptying, increased gastric volume, gastro esophageal reflux, vomiting, aspiration, and VAP. Early and adequate enteral feeding in ICU patients is correlated with decreased overall infections rates, ventilator and intensive care unit (ICU) days, costs, and mortality.

This study is intended to assess the efficacy and safety of the E-Motion System (i.e. E-Motion tubeTM and E-Motion EPG 1000TM) in improving tolerance to enteral nutrition by inducing esophageal motion by means of electrical stimulation in ICU patients.

DETAILED DESCRIPTION:
Malnutrition in the ICU is a known cause for increased morbidity and mortality and providing artificial nutrition is part of standard care in ICUs worldwide. While malnutrition is a risk factor for adverse outcomes related to critical illness, what is more difficult to prove is the value of optimal amounts of nutrition. Nevertheless, large-scale observational studies of critically ill patients suggest that optimal amounts and timely provision of nutritional intake is associated with reduced infectious complications, duration of mechanical ventilation, and mortality, along with perceptions of faster physical recovery. Smaller RCTs demonstrate that greater nutrition intake is associated with improved weaning from mechanical ventilation while larger RCTs do suggest non-significant improvements in long-term physical functional performance (6 minute walk test at 12 months) and a significant improvement in 60-day quality of life. In contrast, there are large-scale RCTs that fail to demonstrate a positive treatment effect of enhanced nutritional intake. However, these trials have been criticized for study heterogeneous groups of low 'nutritional-risk' patients. Patients who benefit the most from optimal nutritional supplementation are high-nutritional risk. Recent data suggests that tolerating 80% of the prescribed amounts of protein and calories is associated with improved clinical outcome and may serve as a quality indicator for ICU practice. Currently, around the world, more than 75% of nutritionally-high risk patients are systematically underfed receiving less than 80% of prescribed amounts. Thus, the investigators conclude that greater efforts to improve nutrition intake in ICU patients are warranted.

Early enteral nutrition (EN) is supported by mechanistic data delineating its physiologic effects, which provide both non-nutritional and nutritional benefits to the critically ill patient. EN should be started as soon as possible following admission to the ICU in order to achieve the non-nutritional benefits and minimize the development of a protein-calorie deficit that frequently occurs during the first week of critical illness. The non-nutritional benefits are derived from several physiologic mechanisms that maintain structural and functional gut integrity, preventing increases in intestinal permeability. Immune mechanisms elicited by EN result in attenuation of oxidative stress and the inflammatory response while supporting the humoral immune system. Enteral feeding modulates metabolic responses that help decrease insulin resistance. The nutritional benefits are derived from delivery of exogenous nutrients, which provide sufficient protein and calories, deliver micronutrients and antioxidants, and maintain lean body mass.

Because many factors impede delivery of early EN in the ICU setting, patients routinely get approximately 50% of the calories and protein that are required. Our mission, at E-Motion Medical, is to improve outcome for critically ill patients by lowering their risk of infection and enabling them to have better nutritional intake. To achieve that, novel technology was developed that reduces gastric reflux and promotes GI motility, via electric stimulation to the esophageal mucosa. The investigators believe our technology will improve gastric emptying, reduce reflux and aspiration of gastric content, and enable more adequate delivery of enteral nutrition to critically-ill patients predisposed to delayed gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-85 years of age.
2. Patient is receiving a moderate to high dose of opioids, either continuously or intermittently and is expected to remain on opioids for an additional 48 hours from point of screening. By moderate to high dose, we mean at least 2 mg/h (or 48 mg/day) of morphine or equivalent (e.g., 20 µg/h fentanyl and 0.5 mg/h of hydromorphone).
3. Mechanically ventilated and expected to remain alive and invasively mechanically ventilated for an additional 48 hours or longer from the point of screening.
4. Receiving EN or prescribed to receive EN.
5. Written informed consent obtained from legal representative (the subject will not be competent to give it on their own).

Exclusion Criteria:

1. Mechanical ventilation start time in your ICU to time of screening is more than 72 hours
2. Subject has a history of or had undergone esophageal or gastric surgery on this admission (lower abdominal surgery will not result in exclusion unless it carries a contraindication to enteral feeding).
3. Subject has a contraindication to enteral feeding (i.e., ongoing bowel obstruction or perforation).
4. Subject requires small bowel feeding at point of screening.
5. Subject requires feeding tube placed operatively or percutaneously.
6. Subject requires total parenteral nutrition at point of screening.
7. Subject has a known diagnosis of gastroparesis requiring outpatient motility agents (e.g. diabetic gastroparesis).
8. Subject has contraindication to oro/nasogastric tube insertion, e.g. esophageal tumors, laryngectomy, etc.
9. Subject with known esophageal varices.
10. Subject has admission diagnosis of gastroesophageal bleeding requiring transfusions.
11. Subject is implanted with a cardiac pacemaker ; temporary pacemaker or is pacemaker dependent ; or implantable defibrillator.
12. Subject has a gastric pacemaker.
13. Subject is prescribed to have NAVA tube or has one in place.
14. Subject is suffering from life-threatening arrhythmia (atrial fibrillation [AF} with rapid ventricular response; sustained VT; ventricular fibrillation [VF]; cardiac arrest; any cardiac arrhythmia that may cause the patient to be hemodynamically instable); severe cardiomyopathy diagnosed clinically or severe congestive heart disease (NYHA 3/4).
15. Subjects with severe hepatic failure (e.g. Child Pugh class C cirrhosis) or acute fulminant hepatic failure. Gilbert's syndrome or asymptomatic gallstones will not result in exclusion.
16. A requirement for continuous EEG monitoring at the time of screening
17. Lactating or pregnant females as determined by positive serum or urine hCG test prior to enrolment.
18. Concomitant participation in another randomized trial of a novel biological or device (non-industry sponsored or academic randomized trials and observational studies are suitable for co-enrolment).
19. Previous randomization in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Adequacy of enteral nutrition | 7 days
  The primary endpoints for this study are the average daily delivery of enteral nutrition in percentage of the amount of calories and protein prescribed for the patient).

SECONDARY OUTCOMES:
Time from intervention start to delivery of 80% prescribed energy and protein | 7 days
  Time (in days) from start of intervention up to delivery of 80% of the calories and/or protein prescribed to the patient in a given day.
Proportion of subjects achieving >80% enteral nutrition intake | 7 days
  Percent of subjects achieving enteral nutrition intake greater than 80% of the amount of calories and/or protein prescribed for the patient each day.

OTHER OUTCOMES:
Pepsin concentration | 7 days
  Pepsin concentration in samples taken daily by ETA (ELISA immunoassay), indicating presence of gastric content in lungs.
microbiological analysis of endotracheal aspirates | 7 days
  Bacterial culture in samples taken daily by ETA.
ICU Length of Stay | 28 days
  Number of days from admission to the ICU until discharge from the ICU.
Pneumonia | 28 days
  Pneumonia infection, as determined by the PI
Ventilator Free Days | 28 days
  Ventilator-free days (number of days alive and free of mechanical ventilation in the first 28 days).
Parenteral Nutrition | 7 days
  Daily delivery of parenteral nutrition calories and/or protein administered.

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit
Locations (11):
- Canada (11):
  - Royal Alexandria Hospital, Edmonton, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences, London, Ontario
  - Ottawa OHRI, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital Sacre-Coeur, Montreal, Quebec
  - Hoptial L'ENfant Jesus, Québec, Quebec
  - University of Sherbrooke Fleurimont, Sherbrooke, Quebec

REFERENCES:
- [Background] Alberda C, Gramlich L, Jones N, Jeejeebhoy K, Day AG, Dhaliwal R, Heyland DK. The relationship between nutritional intake and clinical outcomes in critically ill patients: results of an international multicenter observational study. Intensive Care Med. 2009 Oct;35(10):1728-37. doi: 10.1007/s00134-009-1567-4. Epub 2009 Jul 2. PMID 19572118
- [Background] Heyland DK, Stephens KE, Day AG, McClave SA. The success of enteral nutrition and ICU-acquired infections: a multicenter observational study. Clin Nutr. 2011 Apr;30(2):148-55. doi: 10.1016/j.clnu.2010.09.011. Epub 2010 Oct 25. PMID 20971534
- [Background] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- See also: Sponsor website — http://www.emotionmed.com